CLINICAL TRIAL: NCT04595773
Title: COVID-19, Chronic Adaptation and Response to Exercise (COVID-CARE): A Randomized Controlled Trial
Brief Title: COVID-19, Chronic Adaptation and Response to Exercise (COVID-CARE)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 10000102; 000102-CC
Record Dates: First submitted 2020-10-20; First posted 2020-10-22 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06-10

CONDITIONS: COVID-19
Keywords: Aerobic Exercise Training; Physical Function; Physical Activity; Convalescence; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Motor Activity; Convalescence | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Training and Education (AET+) (Experimental): Participants will perform both exercise training and education for 10 weeks
  Interventions: Other: Aerobic Exercise Training; Other: Education
- Education only (CON) (Other): Participants will perform only education for the first 10 weeks, then cross-over to perform exercise in the second 10 weeks
  Interventions: Other: Aerobic Exercise Training; Other: Education

INTERVENTIONS:
Other: Aerobic Exercise Training — Aerobic exercise training will consist of 10 weeks of aerobic exercise, performed 3 times/week for 30 minutes. Each session will include a warm-up and cool-down period. The intensity will be guided by heart rate and gradually increased from light-moderate to moderate-high intensity as safely tolerated by the subject. All sessions are supervised by credentialed RMD staff members.
Other: Education — Education consisting of weekly lectures lasting approximately 1 hour for 10 weeks. Topics related to exercise programming, safety and well-being will be covered. Conducted remotely by credential RMD staff members.

SUMMARY:
Background:

People who are recovering from COVID-19 may continue to have problems that affect their daily life. For instance, they might feel overly tired. Researchers want to learn if exercise can help people recover after COVID-19 infection.

Objective:

To study if participation in a rehabilitation exercise program can help people recovering from COVID-19.

Eligibility:

Adults ages 18-80 with a lab-confirmed SARS-CoV2 infection (the virus that causes COVID-19), and are still having some symptoms.

Design:

Participants will have a medical history and physical exam. They will give blood and urine samples. They will have tests to measure heart and lung function. Their blood vessels will be assessed.

Participants will have a computed tomography scan of the body. They will have an ultrasound of the muscles in their arms, legs, and chest.

Participants will take a 6-minute walk test. They will take other balance and movement tests.

Participants will walk on a treadmill while hooked up to a monitor. Then they will be interviewed. It will be audio-recorded.

Participants will complete surveys about their symptoms and daily activities.

Participants will take a smell test. For this, they will identify different smells. They will also have memory, attention, and mental functioning tests.

Participants will wear an activity monitor on their wrist 24 hours a day. They will exercise 3 times a week for 10 weeks by moving vigorously on a track or treadmill for 30 minutes. They will attend education classes once a week for 10 weeks.

Participants will be contacted by phone or email every 3 months for 1 year after they complete the exercise part of the study. They will wear an activity monitor for up to 2 weeks.

DETAILED DESCRIPTION:
Study Description:

This randomized controlled trial will determine whether aerobic exercise training has a beneficial effect on physical function, health-related quality of life, free-living physical activity and sleep quality among survivors of COVID-19. Participants will be randomized to either an aerobic exercise training and education (AET+) group or a control education only group (CON) for 10 weeks. Assessments for physical function, self-reported health outcomes for quality of life (QOL), free-living physical activity and sleep quality will be measured at baseline and following the 10-week intervention period. Participants in the CON group will then crossover and perform AET after the 10-week follow-up visit. All participants will be monitored for one year to capture free-living physical activity, sleep quality and health-related QOL outcomes over time. It is hypothesized that following 10 weeks, physical function, health-related QOL, free-living physical activity and sleep quality will show greater improvement with AET+.

Objectives:

Primary Objective:

To examine the effect of aerobic exercise training on physical function in participants recovering from COVID-19.

Secondary Objectives:

To examine the effect of aerobic exercise training on patient reported outcomes and other health-related QOL components in participants recovering from COVID-19; To examine the effect of aerobic exercise training on free-living physical activity and sleep quality in participants recovering from COVID-19.

Exploratory Objectives:

To explore the effect of aerobic exercise training on clinical outcomes, cardiorespiratory function, cognition, biomarkers, metabolomics, ultrasound-based muscle measurements, and vascular function in participants recovering from COVID-19; To explore the feasibility of conducting the AET program remotely in the crossover CON group of participants recovering from COVID-19; To explore follow-up physical activity, sleep quality and health-related QOL outcomes over 1 year in participants recovering from COVID-19.

Endpoints:

Primary Endpoints:

Physical function as measured by distance walked during the 6 minute walk test after 10 weeks post-randomization with AET+ and CON.

Secondary Endpoints:

Patient-reported outcomes and other health-related components after 10 weeks post-randomization with AET+ and CON; Free-living physical activity and sleep quality after 10 weeks post-randomization with AET+ and CON.

Exploratory Endpoints:

Clinical outcomes, cardiorespiratory function, cognition, biomarkers, metabolomics, ultrasound-based muscle measurements, and vascular function after 10 weeks post-randomization with AET+ and CON; Collection of initial feasibility data to conduct exercise sessions remotely; Explore relationships between the physiological variables and post-study health outcome variables over time.

ELIGIBILITY:
* INCLUSION CRITERIA:

Screening procedures will be performed as part of this study. In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Male or female, aged 18 to 80 years
* Previous infection with SARS-CoV2 at least 4 weeks prior to enrollment, confirmed by laboratory or a healthcare provider. Participants with a documented positive home antigen test will need confirmation of positive COVID-19 antibodies (positive anti-Nucleocapsid antibody test, OR positive anti-Spike antibody test if unvaccinated at the time of the antibody test) to be considered.
* Presence of physical limitations or significant fatigue since COVID-19 as demonstrated by:

  * Total score <= 19 on the PROMIS short form for physical function or total score >= 9 on the PROMIS short form for fatigue, AND
  * Score >= 1 on the Patient Global Rating of Flu Severity and Patient Global Assessment of Interference with Daily Activities
* Absence of post-exertional malaise (PEM) as identified on the DSQ-PEM where:

  * Items 1 to 5 has no score >= 2 for frequency and no score >= 2 for severity, occurring in the same row, AND
  * Item 7 or 8 is No , AND
  * Item 9 is <= 13 hours
* Able to read, speak and understand English or Spanish
* Able to understand and willing to sign a written informed consent document
* Willing and able to complete study procedures

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Above normal performance (i.e, >=100% predicted) in the 6MWT based on normative data for gender and age
* History or cardiac condition as determined by NIH cardiology to be unsafe for exercise participation (e.g. ischemic heart disease, right- or left-sided heart failure, cor pulmonale or pulmonary hypertension, dilated or hypertrophic cardiomyopathy or non-idiopathic cardiomyopathy)
* Significant hepatic or renal dysfunction
* Cancer diagnosis with evidence of metastasis or a life expectancy of less than one year
* History of stroke resulting in impairments in functional mobility that limits safe participation
* Active substance abuse including EtOH
* Severe psychiatric disease, not responsive to treatment or medication
* History of diabetes and on insulin pump therapy, or uncontrolled diabetes with HbA1c > 9.0%
* Pregnancy
* Acceptance onto a lung transplant waiting list
* Extreme obesity with BMI > 40 kg/m2
* On medications that would influence exercise performance such as beta blockers or antiretroviral therapy
* Ongoing tobacco and/or nicotine product use
* Enrolled in another interventional clinical research trial
* Any other medical or health condition(s) that unduly increases the risk of exercise testing or training, affects the normal physiologic response to exercise testing or training, and/or would otherwise interfere with the ability to interpret the data as determined by the PI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test distance | Baseline, 10 weeks, 20 weeks (for cross-over group)
  The 6MWT distance has been used to reflect longitudinal changes in physical function among patients with acute lung disease and SARS. A minimal important difference (MID) has yet to be established among survivors of COVID-19. We will consider 30 meters as the MID for this study based on reported ranges of 20 to 30 meters in patients with lung disease.

SECONDARY OUTCOMES:
Patient reported outcomes and quality of life | Baseline, 10 weeks, 20 weeks (for cross-over group), every 3 months for 1 year after exercise
  Patient reported outcomes related to fatigue, sleep, post-traumatic stress disorder, depression, anxiety, general and COVID-19 specific QOL outcomes will be captured.
Free-living physical activity and sleep quality | Baseline, 10 weeks, 20 weeks (for cross-over group), every 3 months for 1 year after exercise
  Quantification of free-living physical activity and sleep quality and patterns using wearable accelerometer device.

CONTACTS AND LOCATIONS:
Overall Officials: Leighton Chan, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000102-CC.html